CLINICAL TRIAL: NCT04555863
Title: haMSter: a Novel Smartphone Communication Tool for People With MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Patrick Altmann MD PhD, Principal Investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1798/2019
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: M-health; Multiple Sclerosis
Keywords: m-health; multiple sclerosis; patient reported outcomes
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- haMSter app (Experimental): Patients receiving the app for personal use for 6 months
  Interventions: Device: haMSter smartphone app

INTERVENTIONS:
Device: haMSter smartphone app — the app tracks patient reported outcomes

SUMMARY:
haMSter is a smartphone app that tracks validated patient reported outcome measures (PROMs) in people multiple sclerosis (MS). In this study, 50 patients with MS will receive this app for 6 months and be asked to fill out the PRO questionnaires on their Smartphone.

Endpoints include the adherence to this app and satisfaction with this Intervention.

ELIGIBILITY:
Inclusion Criteria:

* Any MS according to MacDonald criteria
* informed consent

Exclusion Criteria:

- language barriers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
adherence to device | over the course of this study (over 6 months)
  Percentage (Number) of participants having completed all necessary questionnaires per study period. Max: 6 completions.

SECONDARY OUTCOMES:
Overall satisfaction with this application in telemedicine | after study completion (after 6 months)
  TMPQ (Telemedicine Perception Questionnaire). Min: 0 points. Max: 80 Points. Higher scores indicate a better outcome
General satisfaction with specific Features of the haMSter app | after study completion (after 6 months)
  Empirical questionnaires. We will Report frequencies of answers given. There is no Overall score in a larger sense.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data can only be shared after publication and upon reasonable request made to our local ethics review board.

REFERENCES:
- [Derived] Altmann P, Ponleitner M, Monschein T, Krajnc N, Zulehner G, Zrzavy T, Leutmezer F, Rommer PS, Kornek B, Berger T, Bsteh G. Feasibility of a smartphone app to monitor patient reported outcomes in multiple sclerosis: The haMSter interventional trial. Digit Health. 2022 Nov 4;8:20552076221135387. doi: 10.1177/20552076221135387. eCollection 2022 Jan-Dec. PMID 36353697
- [Derived] Altmann P, Hinterberger W, Leutmezer F, Ponleitner M, Monschein T, Zrzavy T, Zulehner G, Kornek B, Lanzenberger R, Berek K, Rommer PS, Berger T, Bsteh G. The Smartphone App haMSter for Tracking Patient-Reported Outcomes in People With Multiple Sclerosis: Protocol for a Pilot Study. JMIR Res Protoc. 2021 May 7;10(5):e25011. doi: 10.2196/25011. PMID 33960949